CLINICAL TRIAL: NCT02379962
Title: Public Perception and Attitude of Chinese Towards Biomedical Research and Biobank in China
Brief Title: Public Perception and Attitude of Chinese Towards Biomedical Research and Biobanking in China
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yexuan TAO, associate chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2014-087
Record Dates: First submitted 2015-01-26; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Public Knowledge and Attitude Towards Biospecimen-based Research and Their Willingness to Participate in Biobanking
Keywords: biobanking; research participation; China

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
The purpose of this study is to collect date related to public knowledge and attitude towards biospecimen-based research and their willingness to participate in biobanking in China.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18 years and above
* could understand the content of the questionnaire and express themselves
* voluntary to participate in this survey

Exclusion Criteria:

* history of mental illness or the deaf
* not able to express their views and opinions clearly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese people
Sampling Method: Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
measure public knowledge of biobanking and biospecimen-based research with self-complied questionnaire | 4 months
measure public attitude towards biobanking and biospecimen-based research with self-complied questionnaire | 4 months
measure public willingness to participate in biobank with self-complied questionnaire | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- XinHua Hospital Afficilated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China